CLINICAL TRIAL: NCT03559608
Title: Program for the Detection of Hypertension, Its Complications and Factors Predisposing to the Development of Hypertension in Men in the Warmia and Masuria Region
Brief Title: Arterial Hypertension in Men in the Warmia and Masuria Region
Acronym: ProM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Warmia and Mazury (Other)
Collaborators: Zaklady Farmaceutyczne Polpharma SA / Poland (Unknown)
Responsible Party: Principal Investigator, Wojciech Maksymowicz, Head of Collegium Medicum, Clinical Professor, University of Warmia and Mazury
Other Study IDs: ProM
Record Dates: First submitted 2018-04-26; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Arterial Hypertension
Keywords: arterial hypertension; male health; Warmia-Masuria region
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — blood probes and urine probes for laboratory test, frozen samples of serum collected at -80C degree
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to define the prevalence of arterial hypertension and risk factors of its development in an unselected group of Polish men from the region of Warmia and Mazury, considered as one of the most unprivileged in terms of social and employment status in Poland. Polish men life expectancy at birth is 74 years and is lower as polish women life expectancy at birth by 8 years. The difference in Western Europe is 5 years. ProM aims to investigate the prevalence of arterial hypertension as well as to increase the interest in its prevention and treatment in men from the region.

DETAILED DESCRIPTION:
Increased arterial blood pressure (HT) in chronic conditions is a major risk factor of cardiovascular morbidity and premature mortality. HT is diagnosed in 30-45% of global adult population and this number is still growing. The primary aim of the study is to define the prevalence of arterial hypertension and risk factors of its development in an unselected group of Polish men from the region of Warmia and Mazury, considered as one of the most unprivileged in terms of social and employment status in Poland. Polish men life expectancy at birth is 74 years and is lower as polish women life expectancy at birth by 8 years. The difference in Western Europe is 5 years (79 male vs. 84 female) (https://www.statista.com/statistics/274514/life-expectancy-in-europe/).

The study protocol is approved by the Ethics Committee of the Regional Medical Chamber of Warmia and Mazury in Poland. The study are conducted according to the Good Clinical Practice guidelines. Each participant signs an informed consent and be coded with unique ID. As a pivotal part of the ProM project, arterial blood pressure have to be measured in agreement with the ESH/ESC guidelines in randomly selected male subjects. Participants will complete coded and standardized questionnaire and received a referral for free blood and urine tests.

In serum will be tested: glucose, creatinine and lipid profile; microalbuminuria and creatinine were measured in urine, urinary albumin-to-creatinine ratio (UACR) will be calculated. Estimated glomerular filtration rate (eGFR) will be calculated according to the MDRD formula. 1-2 ml of serum will be frozen at -80C degree.

Results of analyses will be saved by indexing with ID code only, personal data with individual IDs will be saved in additional file. All hard copy will be archived in secure room with coded electronic key.

The investigators plan to repeat the measurements in 5 years in follow-up study.

ProM aims to investigate the prevalence of arterial hypertension as well as to increase the interest in its prevention and treatment in men from the region.

ELIGIBILITY:
Inclusion Criteria:

* male

Exclusion Criteria:

* female

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: unselected group of Polish men from the region of Warmia and Mazury
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2022-12-23 (Estimated)

PRIMARY OUTCOMES:
The prevalence of arterial hypertension in men in the region Warmia an Masuria in Poland. | six months after the last inclusion
  For every casual adult male volunteer the arterial blood pressure will be measured in companies, the University, rural areas, stores and markets. Arterial hypertension will be diagnosed in agree with Guidelines ESH/ESC 2013

SECONDARY OUTCOMES:
The prevalence of metabolic syndrom in male population from Warmia and Masuria region in Poland | six months after the last inclusion
  Metabolic syndrome will be diagnosed in participants who will fulfill the criteria of defined by The International Diabetes Federation (2006) and who will participate in free blood tests, waist circumference and blood pressure measurements
Correlation between the parameters measured in blood and arterial blood pressure measurements | six months after the last inclusion
  Sources for the blood parameters will be blood sera collected and frozed at -80C degree from all participants who will participate in free blood tests and blood pressure measurements
The effectiveness of arterial hypertension therapy in men in the region of Warmia an Masuria in Poland | six months after the last inclusion
  All casual volunteers will provide information about the therapy of hypertension in the questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- University Warmia and Mazury, Olsztyn, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Lawes CM, Vander Hoorn S, Rodgers A; International Society of Hypertension. Global burden of blood-pressure-related disease, 2001. Lancet. 2008 May 3;371(9623):1513-8. doi: 10.1016/S0140-6736(08)60655-8. PMID 18456100
- See also: Statistics about life-expectancy-in-europe — https://www.statista.com/statistics/274514/life-expectancy-in-europe/
- See also: Statistics about life-expectancy-in-Poland — http://www.who.int/countries/pol/en/
- See also: IDF consensus 2006 about Metabolic Syndrome — https://web.archive.org/web/20120916064300/http://www.idf.org/webdata/docs/IDF_Meta_def_final.pdf